CLINICAL TRIAL: NCT04407910
Title: Effects of Pre-operative Air-powder Polishing and Rubber-cup Prophylaxis on Tooth Bleaching Outcomes: Randomised Controlled Split-mouth Clinical Study
Brief Title: Office Bleaching Treatment by Using Rubber-cup and Air-powder Polishing Device Prophylaxis in Rondomised Clinical Design
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, zeliha gonca bek kurklu, assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-6-18-78/78
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Tooth Discoloration; Color Changes During Tooth Formation
Keywords: Tooth Bleaching; Prophylaxis; Dental Materials
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: We have two groups applied to split-mouth experimental units. Left side of maxillary have received rubber-cup and right side of maxillary of each subject.have APD prophylaxis respectively.
Who Masked: Participant
Masking Description: Single blind participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air-powder polishing device (Experimental)
  Interventions: Combination Product: AIRFLOW® Master device +Opalescence Xtra Boost.; Combination Product: rubber-cup+Opalescence Xtra Boost.
- Rubber-cup+paste (Experimental)
  Interventions: Combination Product: AIRFLOW® Master device +Opalescence Xtra Boost.; Combination Product: rubber-cup+Opalescence Xtra Boost.

INTERVENTIONS:
Combination Product: AIRFLOW® Master device +Opalescence Xtra Boost. — Prophylaxis techniques for pre-bleaching treatment
Combination Product: rubber-cup+Opalescence Xtra Boost. — Prophylaxis techniques for pre-bleaching treatment

SUMMARY:
The increasing demand for whitening teeth necessitates requirements and guidelines to ensure the efficacy of products and bleaching techniques. So far there is no comparative study to evaluate the effectiveness of pre-operative air-powder polishing device (APD) and rubber-cup prophylaxis on tooth bleaching in-office. Office-bleaching has some advantages such as avoiding soft tissue irritation, preventing the use of excess material and producing immediate esthetic results.

The aim this study is to compare the effects of pre-operative air-powder polishing and rubber-cup prophylaxis on tooth bleaching outcomes. The null hypothesis of this research was that there would be no difference in the change in according to the type of prophylaxis on tooth-bleaching outcomes.△L,△a,△b,△E and △SGU.

The results of the study show that both rubber cup prophylaxis and APD devices can be equally used before bleaching treatment as there were no statistical differences in color change.

DETAILED DESCRIPTION:
Tooth color was measured using spectrophotometer VITA Easyshade V (Vita Zahnfabrik, Germany). The spectrophotometer was calibrated before use in each participant and the device tip was placed on middle thirds of the labial surface of teeth as suggested by the manufacturer's manual.

The tooth color was measured before initial prophylaxis (baseline), immediately after bleaching and after one week. The digital spectrophotometer used in the current study measures the shade of teeth based on the CIE (Commission Internationale de l'éclairage) L*a*b* color space system. This system expresses color as three values: L* for the lightness from black (0) to white (100), a* from green (-) to red (+), and b* from blue (-) to yellow (+). The following values were recorded in the units of CIE L*a*b* color space.

-Data of lightness (L*) and a* and b*axis

-△e: a teeth color change (△e*) was derived as: △e = [(△L *)2+ (△a *)2 + (△b *)2]1/2 While making Shade guide units (SGU) measurements, the bleached index is set according to the VITA Bleached guide 3D-MASTER at spectrophotometer for the measured shade. The measured bleached index after treatment was subtracted from the baseline value. The difference corresponded to the change of the SGU (△ SGU) achieved immediately and 1 week after the bleaching treatment.

The patients had bleaching treatment on the maxillary anterior area including right and left canines. The right and left sides of the patients were randomized by toss of a coin to receive polishing with rubber cup prophylaxis or air powder polishing system before bleaching.

All prophylaxis procedures were performed by same clinician (M.O.). The rubber cup prophylaxis was applied with low-speed handpieces. A rubber cup was attached to the prophy-angle. The handpiece used at a steady slow pace of 2500-3000 rpm. The rubber cup contacted each tooth surface for an average of 5 seconds together with polishing paste consisting of flour of pumice, glycerin and fluoride.

The air polishing treatment was performed by AIRFLOW® Master device (EMS, Nyon, Switzerland) with a six LED (Light Emitting Diode) power setting (2.2 bars dynamic pressure inside powder chamber) and an 11 LED (35 mL/min) water setting for 30 seconds (powder consumption was 1.1 g). Sodium bicarbonate air-powder polishing powder (AIR-FLOW® Plus, EMS Electro Medical Systems, Nyon, Switzerland) was used. The nozzle was held 3-4 mm from the tooth surface and the tip was angulated diagonally. The spray was delivered for an average of 5 seconds using a constant circular motion for each tooth. The spray was directed towards the middle one-thirds of the exposed tooth.

All bleaching procedures were performed by same clinician (Z.G.B.K.). The bleaching agent (Opalescence Xtra Boost/ Ultradent, South Jordan, Utah, USA) was prepared and used following the manufacturer's instructions. Opal Dam (Ultradent, South Jordan, Utah, USA) was used for protection of the gingiva. The bleaching gel was then applied to form 1-2 mm thickness on the buccal surfaces of the teeth of both arches. The gel remained on teeth for 15 minutes and was then suctioned from teeth using a surgical suction tip. This application was repeated a second time in the same session.

ELIGIBILITY:
Inclusion Criteria:

* - being at least 18 years of age
* having minimum of 20 natural teeth (including incisors, canines, and premolars in both arches)
* having good oral hygiene (Plaque index <1, Gingival index <1)

Exclusion Criteria:

* having restorations or active caries on the anterior teeth of either arch
* presence of tetracycline staining or fluorosis
* general hypersensitivity
* gingival recession or periodontal disease
* smokers
* pregnant or lactating women
* history of prior bleaching treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
ΔE | 1 week
  Delta E is a metric for understanding how the human eye perceives color difference

CONTACTS AND LOCATIONS:
Locations (1):
- Zeliha Gonca Bek Kürklü, Adana, Sarıcam, Turkey (Türkiye)

REFERENCES:
- [Background] Sulieman M. An overview of tooth discoloration: extrinsic, intrinsic and internalized stains. Dent Update. 2005 Oct;32(8):463-4, 466-8, 471. doi: 10.12968/denu.2005.32.8.463. PMID 16262034
- [Background] Watts A, Addy M. Tooth discolouration and staining: a review of the literature. Br Dent J. 2001 Mar 24;190(6):309-16. doi: 10.1038/sj.bdj.4800959. PMID 11325156
- [Background] Kihn PW. Vital tooth whitening. Dent Clin North Am. 2007 Apr;51(2):319-31, viii. doi: 10.1016/j.cden.2006.12.001. PMID 17532915
- [Background] Gallagher A, Maggio B, Bowman J, Borden L, Mason S, Felix H. Clinical study to compare two in-office (chairside) whitening systems. J Clin Dent. 2002;13(6):219-24. PMID 12518494
- [Background] Joiner A. The bleaching of teeth: a review of the literature. J Dent. 2006 Aug;34(7):412-9. doi: 10.1016/j.jdent.2006.02.002. Epub 2006 Mar 29. PMID 16569473
- [Background] Seghi RR, Denry I. Effects of external bleaching on indentation and abrasion characteristics of human enamel in vitro. J Dent Res. 1992 Jun;71(6):1340-4. doi: 10.1177/00220345920710061201. PMID 1613185
- [Background] Patil SS, Rakhewar PS, Limaye PS, Chaudhari NP. A comparative evaluation of plaque-removing efficacy of air polishing and rubber-cup, bristle brush with paste polishing on oral hygiene status: A clinical study. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):457-62. doi: 10.4103/2231-0762.167723. PMID 26759798
- [Background] Bernardon JK, Ferrari P, Baratieri LN, Rauber GB. Comparison of treatment time versus patient satisfaction in at-home and in-office tooth bleaching therapy. J Prosthet Dent. 2015 Dec;114(6):826-30. doi: 10.1016/j.prosdent.2015.05.014. Epub 2015 Sep 12. PMID 26372629
- [Background] Sawai MA, Bhardwaj A, Jafri Z, Sultan N, Daing A. Tooth polishing: The current status. J Indian Soc Periodontol. 2015 Jul-Aug;19(4):375-80. doi: 10.4103/0972-124X.154170. PMID 26392683
- [Background] Bernardon JK, Sartori N, Ballarin A, Perdigao J, Lopes GC, Baratieri LN. Clinical performance of vital bleaching techniques. Oper Dent. 2010 Jan-Feb;35(1):3-10. doi: 10.2341/09-008CR. PMID 20166405
- [Background] Chowdhary Z, Mohan R. Efficiency of three different polishing methods on enamel and cementum: A scanning electron microscope study. J Indian Soc Periodontol. 2018 Jan-Feb;22(1):18-24. doi: 10.4103/jisp.jisp_40_17. PMID 29568167
- [Background] Wiegand A, Drebenstedt S, Roos M, Magalhaes AC, Attin T. 12-month color stability of enamel, dentine, and enamel-dentine samples after bleaching. Clin Oral Investig. 2008 Dec;12(4):303-10. doi: 10.1007/s00784-008-0195-7. Epub 2008 Mar 28. PMID 18369668
- [Background] Giachetti L, Bertini F, Bambi C, Nieri M, Scaminaci Russo D. A randomized clinical trial comparing at-home and in-office tooth whitening techniques: A nine-month follow-up. J Am Dent Assoc. 2010 Nov;141(11):1357-64. doi: 10.14219/jada.archive.2010.0081. PMID 21037194
- [Background] Barry TN, Bailey CW, Ashcraft-Olmscheid D, Vandewalle KS. Effect of a New Bleaching Gel on Tooth Whitening. Oper Dent. 2017 Sep/Oct;42(5):559-566. doi: 10.2341/16-200-L. PMID 28829933
- [Background] Nakamura T, Saito O, Ko T, Maruyama T. The effects of polishing and bleaching on the colour of discoloured teeth in vivo. J Oral Rehabil. 2001 Nov;28(11):1080-4. doi: 10.1046/j.1365-2842.2001.00762.x. PMID 11722726
- [Background] Petersilka GJ, Ehmke B, Flemmig TF. Antimicrobial effects of mechanical debridement. Periodontol 2000. 2002;28:56-71. doi: 10.1034/j.1600-0757.2002.280103.x. PMID 12013348
- [Background] Muzzin KB, King TB, Berry CW. Assessing the clinical effectiveness of an aerosol reduction device for the air polisher. J Am Dent Assoc. 1999 Sep;130(9):1354-9. doi: 10.14219/jada.archive.1999.0407. PMID 10492544
- [Background] Goldberg M, Grootveld M, Lynch E. Undesirable and adverse effects of tooth-whitening products: a review. Clin Oral Investig. 2010 Feb;14(1):1-10. doi: 10.1007/s00784-009-0302-4. Epub 2009 Jun 20. PMID 19543926
- [Derived] Kurklu ZGB, Ozcan M. Effects of preoperative air-powder polishing and rubber-cup prophylaxis on tooth bleaching: randomized controlled split-mouth clinical study. Clin Oral Investig. 2021 Oct;25(10):6007-6014. doi: 10.1007/s00784-021-04023-2. Epub 2021 Jun 18. PMID 34145478
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/